CLINICAL TRIAL: NCT04624412
Title: Effects of Different Intensities of Continuous Aerobic Exercises on Fatigue Levels, Mental Well-Being & Mindfulness in Cardiac Rehab Phase 2
Brief Title: Different Intensities of Continuous Aerobic Exercises in Cardiac Rehab Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00711 Mehwish Iftikhar
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Aerobic Moderate Intensity Exercise (Experimental): (Treadmill walking exercise) 50% - 70% of max Heart Rate (HR) (3-6 METS)
  Interventions: Other: Continuous Aerobic Moderate Intensity Exercise
- Continuous Aerobic (Mild intensity Exercise) (Experimental): (Treadmill walking exercise) 30% -50 % of max HR (1-3 METS)
  Interventions: Other: Continuous Aerobic (Mild intensity Exercise)

INTERVENTIONS:
Other: Continuous Aerobic Moderate Intensity Exercise — Continuous Aerobic Moderate Intensity Exercise
  * 5-10 min warm up
  * 30 min moderate aerobic exercise (Treadmill walking exercise)
  * Constant intensity at 50% - 70% of max HR (3-6 METS)
  * 5-10 min cool down
  Arms: Continuous Aerobic Moderate Intensity Exercise
Other: Continuous Aerobic (Mild intensity Exercise) — Continuous Aerobic (Mild intensity Exercise)
  * 5-10 min warm up
  * 30 min mild aerobic exercise (Treadmill walking exercise)
  * Constant intensity at 30-50 % of max HR (1-3 METS)
  * 5-10 min cool down
  Arms: Continuous Aerobic (Mild intensity Exercise)

SUMMARY:
To determine the effects of different intensities of Continuous Aerobic Exercises on Fatigue levels, Mental Well- Being & Mindfulness in Cardiac Rehab Phase 2.

DETAILED DESCRIPTION:
Physical activity has a strong association with health outcomes as it enhances physical and mental function by maximising cardio respiratory fitness and reduces the risk of multiple chronic diseases.

Aerobic exercise is the type of physical activity that accelerates and maintain fitness, well being and quality of life of human being. Aerobic means in presence of oxygen and is based on the power generating process by the utilization of oxygen as a major fuel to cope up the energy demands during sustained physical activity. During Aerobic exercise lungs get more efficient by enhancing their breathing capacity which leads to the removal of carbon dioxide and maximal utilization of oxygen and improvement of its transport to lungs and muscles by circulating blood. Aerobic is the form of exercise which helps in oxygen transportation and absorption while enhancing the efficiency of cardiovascular system. Long term aerobic exercises significantly affect the structure of heart and improve stroke volume of heart.

Fatigue is a feeling of tiredness and leads towards the inability of muscles to perform physically. It is mostly complained during cardiovascular disease and affects the functioning and quality of life in cardiac patients.

Mental well-being is an important constituent of health. Good mental health proves to be beneficial for patients' recovery and independency in activities of daily living. Chronic diseases have a very strong association with mental disorder.

Mindfulness is the ability to be fully alert and mental presence in the moment. Physical training boosts the mindfulness by enhancing the functioning of anterior cingulate cortex that has been linked to the improvement of self-regulation and attention. Aerobic exercises can improve the mood mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) (class 1, class II)
* Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
* Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
* Post Coronary artery bypass grafting (CABG)
* Patients diagnosed with mild to moderate depression on basis of Patient Health Questionnaire (PHQ-9)

Exclusion Criteria:

* Recurrent myocardial ischemia or Infarction (MI)
* Unstable angina
* Any diagnosed psychological disease
* Patients with impaired cognition function
* Patients with severe life-limiting illness such as cancer, and renal failure.
* Congestive Heart failure

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Borg Scale Rate of Perceived Exertion | 6th week
  Changes from the Baseline will be measured, This scale is from 6-20 , where 6 means no exertion at all and 20 means maximal exertion, A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.
Fatigue Severity Scale | 6th week
  Changes from the Baseline will be measured, The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders. A self-report scale of nine items about fatigue, its severity and how it affects certain activities. Answers are scored on a seven-point scale where 1 = strongly disagree and 7 = strongly agree. This means the minimum score possible is nine and the highest is 63.
Mindfulness attention awareness scale | 6th week
  Changes from the Baseline will be measured, The trait Mindfulness attention awareness scale (MAAS) is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place. To score the scale simply compute the mean of the fifteen items. Higher scores reflect higher levels of dispositional mindfulness.
The Warwick Edinburgh mental Well- being scale | 6th week
  Changes from the Baseline will be measured, The Warwick-Edinburgh Mental Well being Scales (WEMWBS) were developed to enable the measuring of mental wellbeing in the general population and the evaluation of projects, programmes and policies which aim to improve mental well-being. The 14-item scale WEMWBS has 5 response categories, summed to provide a single score. The items are all worded positively and cover both feeling and functioning aspects of mental well-being, thereby making the concept more accessible. The scale has been widely used nationally and internationally for monitoring, evaluating projects and programmes and investigating the determinants of mental wellbeing. The minimum scale score is 14 and maximum is 70. The scale is scored by summing responses to each item answered on a 1 to 5 likert scale.
Patient Health Questionnaire | 6th week
  The Patient Health Questionnaire (PHQ-9) is the depression module, which scores each of the nine Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria as "0" (not at all) to "3" (nearly every day). It has been validated for use in primary care. It is not a screening tool for depression but it is used to monitor the severity of depression and response to treatment. However, it can be used to make a tentative diagnosis of depression in at-risk populations - those with coronary heart disease or after stroke.
Ejection fraction | 6th week
  Changes from the Baseline will be measured, Echocardiography is a test that uses sound waves to produce live images of your heart. The image is an echocardiogram. This test allows your doctor to monitor how your heart and its valves are functioning. Ejection fraction (EF) is a measurement of the percentage of blood leaving your heart each time it contracts. The heart contracts and relaxes. A normal heart's ejection fraction may be between 50 and 70 percent. A ejection fraction measurement under 40 percent may be evidence of heart failure or cardiomyopathy. EF from 41 to 49 percent may be considered "borderline." It does not always indicate that a person is developing heart failure. Instead, it may indicate damage, perhaps from a previous heart attack. An ejection fraction measurement higher than 75 percent may indicate a heart condition such as hypertrophic cardiomyopathy.
6 min walk test: Distance (meters) | 6th week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min without any support.
Pulse Rate | 6th week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter
Oxygen Saturation (SpO2) | 6th week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Systolic and diastolic blood pressure | 6th week
  Changes from the Baseline, Blood pressure is measured through sphygmomanometer
Multidimensional assessment of fatigue | 6th week
  Changes from the Baseline, The Multidimensional assessment of fatigue (MAF) is a 16 item scale that measures fatigue according to four dimensions: degree and severity, distress that it causes, timing of fatigue (over the past week, when it occurred and any changes), and its impact on various activities of daily living (household chores, cooking, bathing, dressing, working, socializing, sexual activity, leisure and recreation, shopping, walking, and exercising). Numerical rating scale (1 - 10) for items 1, and 4 - 14 ( 1 = not at all, 10 = a great deal), item 2 (1 = mild to 10 = severe), item 3 ( 1 = no distress, 10 = a great deal of distress). Categorical responses (1 - 4) for Timing items 15 and 16. A higher score indicates more severe fatigue, fatigue distress, or impact on activities of daily living.
Lipid Profile test | 6th week
  Changes from the Baseline was measure after taking blood samples, Lipid Profile test includes following: Low-density lipoprotein cholesterol (LDL-C) at goal (<100mg/dL), high-density lipoprotein cholesterol (HDL-C) within normal range (40mg/dL for males and 50mg/dL for females), and/or triglycerides within normal range (≤ 150mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSPT-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Rawalpindi Institute of Cardiology, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No